CLINICAL TRIAL: NCT03841903
Title: Structural Analysis of Spinal Cord Grey and White Matter Changes in Patients With Multiple Sclerosis: Sub-study Within the Swiss Multiple Sclerosis Cohort (SMSC-study)
Brief Title: Spinal Cord Analysis in Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-01461; me16Kappos2
Record Dates: First submitted 2019-02-11; First posted 2019-02-15 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Multiple Sclerosis
Keywords: Spinal cord; Spinal cord atrophy; Cerebrospinal Fluid; Swiss Multiple Sclerosis Cohort
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- relapsing-remitting MS undergoing spinal cord MRI
  Interventions: Diagnostic Test: spinal cord MRI
- secondary progressive MS undergoing spinal cord MRI
  Interventions: Diagnostic Test: spinal cord MRI
- primary progressive MS undergoing spinal cord MRI
  Interventions: Diagnostic Test: spinal cord MRI
- healthy control (HC) undergoing spinal cord MRI
  Interventions: Diagnostic Test: spinal cord MRI

INTERVENTIONS:
Diagnostic Test: spinal cord MRI — high-resolution spinal cord MRI sequences on a 3Tesla magnet (Siemens Prisma) with high contrast between SC and CSF as well as high contrast within the SC (grey-white matter contrast)

SUMMARY:
Research project in which patients with Multiple Sclerosis (MS) are examined clinically and with magnetic resonance imaging (MRI). To evaluate spinal cord (SC) grey and white matter changes (incl. lesions) using fast, high-resolution MRI sequences with high contrast between SC and cerebrospinal fluid (CSF) as well as high contrast within the SC (grey-white matter contrast).

DETAILED DESCRIPTION:
The Swiss Multiple Sclerosis Cohort (SMSC-Study) aims to better evaluate specific Multiple Sclerosis (MS) phenotypes through the systematic and standardised documentation and acquisition of clinical course and paraclinical tests such as magnetic resonance imaging (MRI), blood and cerebrospinal fluid (CSF) specimens.

Determination of the relative contribution of SC metrics (cervical cord volume, cervical grey matter (GM) cord volume, cervical white matter (WM) cord volume, SC lesion load) to disability in MS.

ELIGIBILITY:
Inclusion criteria

* Diagnosis of multiple sclerosis
* Steroid free period: > 4 weeks
* healthy controls without any history of severe neurological, internistic or psychiatric disease

Exclusion Criteria for all participants:

* History of severe (other) neurological, internistic or psychiatric disease
* MRI related exclusion criteria:

  1. Paramagnetic and/or superparamagnetic foreign objects in the body
  2. Pacemaker
  3. Claustrophobia
  4. Pregnancy, lactation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The recruitment of MS patients will take place within the ongoing SMSC study at the MS Clinic of the Department of Neurology (Neurologische Klinik und Poliklinik), University Hospital Basel (Universitätsspital Basel). Healthy subjects will be recruited by public announcements on the University Hospital's and the University's notice board.
Sampling Method: Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2020-03-24 (Actual); Study Completion 2020-03-24 (Actual)

PRIMARY OUTCOMES:
Change in SC atrophy assessed by MRI | at baseline and after 1 year
  Determination of the degree of SC grey and white matter atrophy in MS patients with relapsing versus progressive disease courses in comparison to matched HC. Measurement tool is a structural MRI of the brain and spinal cord at 3 Tesla. Assessment will last approx. 90 minutes.

SECONDARY OUTCOMES:
Change in Timed 25-foot walk test (T25-FW) | at baseline and after 1 year and after 5 years
  Quantitative mobility and leg function performance test ( in MS patients) based on a timed 25-walk. The patient is directed to one end of a clearly marked 25-foot course and is instructed to walk 25 feet as quickly as possible, but safely. The time is calculated from the initiation of the instruction to start and ends when the patient has reached the 25-foot mark.
Change in Multiple Sclerosis Walking Scale-12 (MSWS-12) Questionnaire | at baseline and after 1 year and after 5 years
  Self-assessment scale which measures the impact of MS on walking. It consists of 12 questions concerning the limitations to walking due to MS during the past 2 weeks. Each item can be answered with 5 options, with 1 meaning no limitation and 5 extreme limitation.

CONTACTS AND LOCATIONS:
Overall Officials: Ludwig Kappos, Prof. Dr. MD, Principal Investigator — Department of Neurology University Hospital Basel
Locations (1):
- Dep. of Neurology, University Hospital Basel, Basel, Switzerland